CLINICAL TRIAL: NCT07024303
Title: Measuring the Effects of Medication and Behavioral Treatments for Challenging Behavior
Brief Title: Measurement of Treatment Effects
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Matthew J O'Brien, PhD, BCBA-D (Other)
Responsible Party: Sponsor-Investigator, Matthew J O'Brien, PhD, BCBA-D, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202411526
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Challenging Behavior; Autism Spectrum Disorder
Keywords: psychotropic medication; behavioral therapy; behavioral measurement
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: This is a non-randomized (preference) parallel group design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Psychotropic Medication (Experimental): Classes of psychotropic medications used as treatment for challenging behavior include antipsychotics (e.g., aripiprazole, quetiapine), stimulants (e.g., methylphenidate), alpha 2 agonists (e.g., clonidine), and mood-stabilizing anticonvulsants (e.g., valproate). However, other classes of psychotropics may be used to indirectly address challenging behavior (e.g., anxiolytics, antidepressants). Two medications (aripiprazole and risperidone) are FDA approved to treatment irritability for individuals with autism and challenging behavior. Psychotropic medications range in timing and dosage and their effects may be immediate (e.g., stimulants) or take as long as 6 weeks for full therapeutic effects (e.g., risperidone).
  Interventions: Drug: Psychotropic medication (at discretion of psychiatrist)
- Behavior Therapy (Experimental): In this study, FCT treatment will be provided weekly for approximately 60 min in duration. To facilitate communication during FCT, a word/picture card or microswitch (with recorded voice output) will be paired with any pre-existing child requests. Appropriate requests will be reinforced by the caregiver or therapist, and the occurrence of challenging behavior will be ignored (placed on extinction) or result in the caregiver/therapist providing guided compliance. An individualized FCT treatment plan will be developed based on the results of the functional analysis. For example, if the functional analysis identifies challenging behavior that functioned to escape task demands, then the FCT treatment plan will focus on teaching the child to request breaks appropriately after complying with instructions to complete a task. A typical task demand will be initiated by placing a small amount of developmentally appropriate "work" in front of the child and asking him or her to complete the task
  Interventions: Behavioral: Behavioral therapy
- Combined Treatment (Medication+Behavior Therapy) (Experimental): Participants in this arm will receive both medication and behavior therapy using the same manipulations as the Psychotropic Medication and Behavior Therapy Arms.
  Interventions: Drug: Psychotropic medication (at discretion of psychiatrist); Behavioral: Behavioral therapy
- No Treatment (No Intervention): Participants who chose none of the treatment arms may participate in the assessments.

INTERVENTIONS:
Drug: Psychotropic medication (at discretion of psychiatrist) — The timing and dose of medication will be determined by the prescribing provider. Most medications are delivered daily and some medications may be delivered more than once per day. Providers are expected to adhere to professional guidelines for prescribing.
  Arms: Combined Treatment (Medication+Behavior Therapy); Psychotropic Medication
Behavioral: Behavioral therapy — Functional communication training (FCT) will be delivered for 1 hour every week in-vivo or via telehealth. This timing and dosage has been shown effective in previous research. However, caregivers will be encouraged to practice the treatment procedures as often as possible on their own. Treatment will be delivered by a therapist and/or caregiver for those receiving in-vivo therapy and caregivers will deliver treatment with coaching from a therapist when using telehealth.
  Arms: Behavior Therapy; Combined Treatment (Medication+Behavior Therapy)

SUMMARY:
The overall objective is to evaluate and compare the efficacy of two common treatments for CB in children and adolescents with autism using multiple outcome measures. Our central hypothesis is that both behavioral treatment and medication will produce reductions in CB, but behavioral treatments, including behavior treatment + medication, will produce a greater reduction in CB when measured using direct observation within the contexts most associated with challenging behavior. We have four aims: Aim 1: Evaluate the concordance between indirect and direct measures of challenging behavior. We hypothesize that behavior change (% change) will be discordant between indirect and direct measurement data, regardless of treatment type, with direct measurement resulting in significantly greater change at each measurement timepoint. Aim 2: Compare the efficacy of psychotropic medication, behavior therapy, and combination therapy (medication+behavior therapy) on CB using indirect measures (ABC-I, BPI, CGI, MOSES) and direct observation (antecedent analysis). We hypothesize that all treatment modalities will reduce CB on both outcome measures at each standard timepoint, but behavioral therapy and combination therapy will produce a significantly greater reduction on direct observation of CB in the contexts most associated with challenging behavior. Aim 3: Compare the social validity of psychotropic medication, behavior therapy, and combination therapy using the Treatment Acceptability Rating Form-Revised (Reimers et al., 1992). Aim 4: Compare the social validity of measurement methods (indirect vs. direct).

DETAILED DESCRIPTION:
Our overall objective of this study is to evaluate and compare the efficacy of two common treatments for CB in children and adolescents with autism using multiple outcome measures. Our central hypothesis is that behavioral treatment, medication, and combination treatment (medication+behavior therapy) will produce reductions in CB, but behavioral treatment and combination treatment will produce a greater reduction in CB when measured using direct observation within the contexts most associated with challenging behavior.

To address this objective, we plan to recruit up to 20 individuals under 13 years of age who are diagnosed with autism and exhibit challenging behavior to participate in this study. Subjects will be recruited from clinics where patients receive consultation on medication for challenging behavior. Subjects will be given the options of initiating/continuing medication, initiating behavior therapy, both medication and behavior therapy, or neither medication nor behavior therapy. The behavioral treatment provided as part of the research study will be functional communication training or FCT. FCT is a scientifically validated behavior therapy that involves teaching the child to use communication (in various forms) instead of challenging behavior to get what they want. It will be delivered at a timing (1 time per week) and dosage (60 minutes per visit) that is common for individuals with challenging behavior. Subjects will participate in a baseline behavioral assessment (baseline), as well as monthly behavioral assessments. Each behavioral assessment will include indirect (rating scales) and direct (antecedent analysis) measures of challenging behavior, as well as measures of social validity (treatment acceptability rating scales). Subjects will be followed for 6 months and comparisons of behavior change across measures will be used to determine treatment effectiveness and concordance between measures.

ELIGIBILITY:
The adult subjects will be the caregiver/guardian of the minor subjects. The only inclusion criterion for the adult subjects is that they must be the caregiver/legal guardian of the minor subject and their home is primarily English speaking.

The minor subjects will be individuals who were referred to Child and Adolescent Psychiatry at University of Iowa Healthcare for management of challenging behavior (e.g., physical aggression, self-injury, destruction, elopement, generalized refusal) and meet the following criteria:

1. Between the ages of 2 years, 0 months and 12 years, 0 months
2. Diagnosed with autism spectrum disorder
3. Diagnosed with intellectual disability at the moderate, severe, or profound range (called "profound autism").
4. Display challenging behavior, including one or more of the following: physical aggression, self-injury, destruction, elopement, generalized refusal
5. Live in a home where English is the primary language spoken.
6. The caregiver is considering medication, behavioral therapy, or both to treat the child's challenging behavior.

Subjects would be excluded if:

1. Not diagnosed with autism spectrum disorder
2. Do not have a moderate or severe/profound intellectual disability
3. Do not display challenging behavior
4. Live in a home where English is not the primary language spoken
5. Caregivers are not considering medication, behavior therapy, or both to treat challenging behavior

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist, Irritability Subscale | At enrollment and monthly for 12 months.
  The ABC-I is a subscale of the 58-item ABC rating scale, which more broadly measures irritability, social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech (Aman et al., 1985). Items are rated on a 4-point. Likert scale from 0 to 3, with higher ratings corresponding to greater concern. Recent research has provided normative data for children with ASD, illustrating the validity of the five-factor structure and appropriate convergent and divergent validity (Kaat et al., 2014) as well as excellent internal consistency for the subscale of interest (Irritability = 0.92; Norris et al., 2019). The ABC-I consists of 15 items that measure child irritable mood and is commonly used to measure the effects of pharmacotherapy or behavioral therapy on disruptive behavior in children with autism (Bearss et al., 2015; Goel et al., 2018).
Behavior Problems Inventory | At enrollment and monthly for 12 months.
  The BPI is a 52-item scale used to assess problem behavior in individuals with neurodevelopmental disabilities (Rojahn et al., 2001). Specific behaviors (e.g., hits others, bites self) are scored on a 5-point frequency scale (0 = never, 4 = hourly) and a 4-point severity scale (0 = no problem, 3 = severe problem). The BPI measures three types of behavior: self-injurious behaviors, stereotyped behavior, and aggressive or destructive behavior. The BPI has been determined to demonstrate reasonable validity and reliability (e.g., Rojahn et al., 2001).
Clinical Global Impressions Scale | At enrollment and every month for 12 months.
  The CGI is a comprehensive, clinician-determined summary measure that integrates all available information, including the patient's history, psychosocial context, symptoms, behavior, and the impact of symptoms on functional ability. The CGI consists of two single-item measures: (a) the severity of psychopathology, rated on a 1 to 7 scale, and (b) the change from the initiation of treatment, also rated on a seven-point scale. This measure is delivered following a clinical evaluation. The CGI has shown strong correlations with established research drug efficacy scales. The standard CGI is widely used in FDA-regulated trials.
Home Situations Questionnaire | At enrollment and monthly for 12 months.
  The HSQ-PDD is a 25-item scale used to assess behavioral compliance in everyday settings. It is typically completed by parents of individuals with ASD (Chowdhury et al., 2010). The HSQ-PDD is a modified version of the original HSQ (Barkley & Edelbrock 1987) and includes additional items identified as relevant to children with ASD (e.g., when asked to move from one activity to another; when there is an unexpected change in routine). When completing the measure, the rater must first identify whether an item is a challenge for the child and then rate the severity of the problem on a 9-point Likert scale (1 = mild, 9 = severe). The HSQ-PDD consists of two factors (Socially Inflexible, 14 items; Demand-Specific, 6 items). Internal consistency for the scale as a whole is excellent (Chowdhury et al., 2010).
Monitoring of Side Effects Scale | At enrollment and monthly for 12 months.
  The MOSES will be administered monthly and at the 6-month follow up to evaluate side effects from behavior therapy, medication, or both. The MOSES is a comprehensive caregiver/self-administered rating scale of the potential adverse effects from psychotropic medications. It includes 83 possible symptoms that may affect 8 areas of bodily functioning. It integrates self-report and observational methods. The MOSES was developed based on reviews of psychotropic medications. Items are scored based on a zero (not present) to 4 (severe) scoring system.
Treatment Acceptability Rating Form - Revised | Monthly for 12 months.
  The TARF-R will be administered monthly and at the 6-month follow up. It is a measure of social validity that is often used to evaluate behavioral therapies. The TARF-R consists of 20 items that are rated on a 7-point Likert-type scale: 17 items pertain to caregiver ratings of the total acceptability of the treatment, 2 items to caregiver perception of problem severity for the child, and 1 item to caregiver understanding of proposed intervention.

IPD SHARING:
Plan to Share IPD: No